CLINICAL TRIAL: NCT00073034
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of 3 Fixed Doses of EAA-090 in Adult Outpatients With Neuropathic Pain Associated With Diabetic Neuropathy
Brief Title: Study Evaluating EAA-090 in Adult Outpatients With Neuropathic Pain Associated With Diabetic Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0912A2-212
Record Dates: First submitted 2003-11-14; First posted 2003-11-18 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathy, Painful
Keywords: Neuropathic Pain; Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Neuralgia | interventions — EAA-090

INTERVENTIONS:
Drug: EAA-090

SUMMARY:
EAA-090 is being developed for the treatment of neuropathic pain associated with diabetic neuropathy. It is a selective antagonist that binds competitively to the glutamate site of the N-methyl-D-aspartate (NMDA) receptor.

This study will assess the safety and efficacy of 3 fixed oral doses of EAA-090 compared with placebo in subjects with neuropathic pain associated with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must have a negative serum pregnancy test result at screening
* Diabetes mellitus (type I or II) that is controlled by oral or parenteral hypoglycemic agents or diet
* Diagnosis of painful diabetic distal symmetric sensory/motor polyneuropathy

Exclusion Criteria:

* Pregnancy, lactation, or plans to become pregnant during the study
* Depo-Provera or oral contraceptives that have been taken for less than 1 month before study day 1 if not using another medically accepted form of birth control
* History of multiple drug allergies that may put the subject at greater risk during study participation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer